CLINICAL TRIAL: NCT06246630
Title: A Prospective, Exploratory Study Evaluating the Effectiveness of Treatment Regimens for Locally Advanced/Metastatic Non-resectable Pancreatic Neuroendocrine Tumor (PNET) Guided by in Vitro Drug Sensitivity Testing of Tumor Organoids
Brief Title: In Vitro Organoid Drug Sensitivity-Guided Treatment for Advanced Pancreatic Neuroendocrine Tumor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Chongqing Kingbiotech Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, JIABIN JIN, Associate Chief Physician, Pancreatic Disease Center, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ruijin20231007060328844
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Advanced Pancreatic Neuroendocrine Tumor
Keywords: p-NET; organoid; chemotherapy; target therapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organoid-Guided therapy (Experimental): All patients will be included in a single-arm. Participants will undergo biopsy of tumor tissue for subsequent organoid generation and drug sensitivity tests.
  Interventions: Other: Chemotherapy and targeted-therapy guided by organoid drug sensitivity test

INTERVENTIONS:
Other: Chemotherapy and targeted-therapy guided by organoid drug sensitivity test — this study conducts drug sensitivity tests on various clinically approved drugs. The most sensitive drug for the patient is selected for treatment, and the study aims to evaluate the clinical effectiveness of the drug and its consistency with in vitro organoid drug sensitivity.

SUMMARY:
The purpose of this study is to explore whether chemotherapy and targeted-therapy regimens guided by organoid drug sensitivity test can improve the outcomes of non-resectable locally advanced and metastatic Pancreatic neuroendocrine tumors. At the same time, this study will evaluate the successful stablishment rate of organoid from biopsy tissue , and explore the concordance between drug sensitivity test results and patients' treatment response

DETAILED DESCRIPTION:
Twenty non-resectable locally advanced and metastatic pancreatic neuroendocrine Tumor(p-NET) patients who should receive palliative treatment will be enrolled in this study. Baseline information of the enrolled patients including medical history, physical examination records and clinical examination records will be collected. Tumor material of those patients will be obtained from Pancreatic endoscopic biopsies or surgical resection. Patient-derived organoids (PDOs) will be established and cultured from p-NET tumor specimens. PDOs will then be treated with drugs of the chemotherapeutic and targeted therapeutic regimens for p-NET. Organoid size and growth will be monitored before and after the treatment, and dose-response curves will be generated. As for the assessment of clinical outcomes of patients, treatment responses will be assessed by biomedical imaging according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1). Consistency between treatment responses in PDO models and clinical outcomes of patients will be assessed by correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years old.
2. Histologically or cytologically confirmed locally advanced/metastatic Pancreatic Neuroendocrine Tumor
3. Surgery was considered impossible or can not receive the radical purpose.
4. Able to provide fresh tumor tissue specimens for organoid culture, including: tumor biopsy tissues, tumor surgical specimens, etcy.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2.
6. Expected survival time≥ six months.
7. Patient have been informed and consented, compliance and geographic proximity to ensure adequate follow-up

Exclusion Criteria:

1. Other malignancies in the past 5 years, excluding cured basal cell carcinoma of the skin.
2. History of severe cardiovascular events and myocardial Infarction within twelve months before the study.
3. Patients with psychiatric disorders or with psychotropic substance abuse and inability to abstain.
4. Pregnant or breastfeeding women.
5. According to researcher's consideration, patients with other serious systemic diseases or other conditions that are not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1-2 years
  Percentage of patient's measurable disease who have achieved either complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progressive free survival | 1-2 years
  The time from initiation of treatment to the occurrence of disease progression or death.
Overall survival time | 2 years
  The time from the date of randomization to the date of death for any cause. Patients will be followed until their date of death or until final database closure.
The successful establishment rate of organoids | 1-2 years
  The rate of organoid successfully cultured in all the samples collected.
Concordance between drug sensitivity test results and patients' treatment response | 1-2 years
  To assess the accuracy of drug sensitivity test in both group. The number of patients with correct prediction of treatment response by organoid drug-sensitivity test divided by the number of patients underwent chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jiabin JIN, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 中国临床肿瘤学会神经内分泌肿瘤专家委员会. 中国胃肠胰神经内分泌肿瘤专家共识（2022年版）[J]. 中华肿瘤杂志, 2022, 44(12):1305-1329
- [Background] 吴文铭, 陈洁, 白春梅等.中国胰腺神经内分泌肿瘤诊疗指南（2020） [J] . 中华外科杂志, 2021, 59(6) : 401-421
- [Background] 王文权, 楼文晖, 刘亮.胰腺神经内分泌肿瘤热点问题的思考[J]. 中华消化外科杂志, 2022, 21(8):1031-1037
- [Background] Ribeiro-Filho AC, Levy D, Ruiz JLM, Mantovani MDC, Bydlowski SP. Traditional and Advanced Cell Cultures in Hematopoietic Stem Cell Studies. Cells. 2019 Dec 12;8(12):1628. doi: 10.3390/cells8121628. PMID 31842488
- [Background] Hidalgo M, Amant F, Biankin AV, Budinska E, Byrne AT, Caldas C, Clarke RB, de Jong S, Jonkers J, Maelandsmo GM, Roman-Roman S, Seoane J, Trusolino L, Villanueva A. Patient-derived xenograft models: an emerging platform for translational cancer research. Cancer Discov. 2014 Sep;4(9):998-1013. doi: 10.1158/2159-8290.CD-14-0001. Epub 2014 Jul 15. PMID 25185190
- [Background] Li M, Izpisua Belmonte JC. Organoids - Preclinical Models of Human Disease. N Engl J Med. 2019 Feb 7;380(6):569-579. doi: 10.1056/NEJMra1806175. No abstract available. PMID 30726695
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Background] Yan HHN, Siu HC, Law S, Ho SL, Yue SSK, Tsui WY, Chan D, Chan AS, Ma S, Lam KO, Bartfeld S, Man AHY, Lee BCH, Chan ASY, Wong JWH, Cheng PSW, Chan AKW, Zhang J, Shi J, Fan X, Kwong DLW, Mak TW, Yuen ST, Clevers H, Leung SY. A Comprehensive Human Gastric Cancer Organoid Biobank Captures Tumor Subtype Heterogeneity and Enables Therapeutic Screening. Cell Stem Cell. 2018 Dec 6;23(6):882-897.e11. doi: 10.1016/j.stem.2018.09.016. Epub 2018 Oct 18. PMID 30344100
- [Background] Sharick JT, Walsh CM, Sprackling CM, Pasch CA, Pham DL, Esbona K, Choudhary A, Garcia-Valera R, Burkard ME, McGregor SM, Matkowskyj KA, Parikh AA, Meszoely IM, Kelley MC, Tsai S, Deming DA, Skala MC. Metabolic Heterogeneity in Patient Tumor-Derived Organoids by Primary Site and Drug Treatment. Front Oncol. 2020 May 15;10:553. doi: 10.3389/fonc.2020.00553. eCollection 2020. PMID 32500020
- [Background] Kopper O, de Witte CJ, Lohmussaar K, Valle-Inclan JE, Hami N, Kester L, Balgobind AV, Korving J, Proost N, Begthel H, van Wijk LM, Revilla SA, Theeuwsen R, van de Ven M, van Roosmalen MJ, Ponsioen B, Ho VWH, Neel BG, Bosse T, Gaarenstroom KN, Vrieling H, Vreeswijk MPG, van Diest PJ, Witteveen PO, Jonges T, Bos JL, van Oudenaarden A, Zweemer RP, Snippert HJG, Kloosterman WP, Clevers H. An organoid platform for ovarian cancer captures intra- and interpatient heterogeneity. Nat Med. 2019 May;25(5):838-849. doi: 10.1038/s41591-019-0422-6. Epub 2019 Apr 22. PMID 31011202
- [Background] Shi X, Li Y, Yuan Q, Tang S, Guo S, Zhang Y, He J, Zhang X, Han M, Liu Z, Zhu Y, Gao S, Wang H, Xu X, Zheng K, Jing W, Chen L, Wang Y, Jin G, Gao D. Integrated profiling of human pancreatic cancer organoids reveals chromatin accessibility features associated with drug sensitivity. Nat Commun. 2022 Apr 21;13(1):2169. doi: 10.1038/s41467-022-29857-6. PMID 35449156
- [Background] Dijkstra KK, van den Berg JG, Weeber F, van de Haar J, Velds A, Kaing S, Peters DDGC, Eskens FALM, de Groot DA, Tesselaar MET, Voest EE. Patient-Derived Organoid Models of Human Neuroendocrine Carcinoma. Front Endocrinol (Lausanne). 2021 Mar 11;12:627819. doi: 10.3389/fendo.2021.627819. eCollection 2021. PMID 33776923
- [Background] Kawasaki K, Toshimitsu K, Matano M, Fujita M, Fujii M, Togasaki K, Ebisudani T, Shimokawa M, Takano A, Takahashi S, Ohta Y, Nanki K, Igarashi R, Ishimaru K, Ishida H, Sukawa Y, Sugimoto S, Saito Y, Maejima K, Sasagawa S, Lee H, Kim HG, Ha K, Hamamoto J, Fukunaga K, Maekawa A, Tanabe M, Ishihara S, Hamamoto Y, Yasuda H, Sekine S, Kudo A, Kitagawa Y, Kanai T, Nakagawa H, Sato T. An Organoid Biobank of Neuroendocrine Neoplasms Enables Genotype-Phenotype Mapping. Cell. 2020 Nov 25;183(5):1420-1435.e21. doi: 10.1016/j.cell.2020.10.023. Epub 2020 Nov 6. PMID 33159857